

## **Statistical Analysis Plan**

The Efficacy of MEDIHONEY® for Chronic Rhinosinusitis With Nasal Polyposis After Functional Endoscopic Sinus Surgery NCT02562924
ID: CHRMS 15-010

Original Date: November 19, 2018 Date Updated\*: September 25, 2019 \*Original document date added per request

Baseline comparisons of the 3 study arms used Fisher's exact test for categorical variables and analysis of variance for continuous variables. The arms were compared on changes in the outcome measures from baseline to Day 119 using analysis of variance. No adjustments were made for testing multiple variables since a global null hypothesis was not of interest.

Rothman KJ. No adjustments are needed for multiple comparisons. Epidemiology 1990; 1:43-46.

Perneger TV. What's wrong with Bonferroni adjustments. BMJ 1998; 316:1236-1238